CLINICAL TRIAL: NCT03064854
Title: Phase Ib, Multicenter, Open Label Study of PDR001 in Combination With Platinum Doublet Chemotherapy and Other Immunooncology Agents in PD-L1 Unselected, Metastatic NSCLS Patients (ElevatION:NSCLC-101 Trial)
Brief Title: PDR001 in Combination With Platinum-doublet Chemotherapy and Other Immunology Agents in PD-L1 Unselected, Metastatic NSCLC Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment halted prematurely due to competitive landscape for lung cancer therapies
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPDR001C2101; 2016-002815-17 (EudraCT Number)
Record Dates: First submitted 2017-02-06; First posted 2017-02-27 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PDR001; immunotherapy; Non-small cell lung cancer; lung; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — spartalizumab; Cisplatin; Gemcitabine; Pemetrexed; Carboplatin; Paclitaxel; canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A: squamous, gem/cis+PDR001 (Experimental)
  Interventions: Drug: PDR001; Drug: Cisplatin; Drug: Gemcitabine
- Group B: non-squamous, pem/cis+PDR001 (Experimental)
  Interventions: Drug: PDR001; Drug: Cisplatin; Drug: Pemetrexed
- Group C: paclitaxel/carbo+PDR001 (Experimental)
  Interventions: Drug: PDR001; Drug: Carboplatin; Drug: Paclitaxel
- Group E: non-squamous, pem/cis (or carbo)+PDR001+canakinumab (Experimental)
  Interventions: Drug: PDR001; Drug: Cisplatin; Drug: Pemetrexed; Drug: Carboplatin; Drug: Canakinumab

INTERVENTIONS:
Drug: PDR001 — Powder for solution for infusion
Drug: Cisplatin — Intravenous infusion
  Arms: Group A: squamous, gem/cis+PDR001; Group B: non-squamous, pem/cis+PDR001; Group E: non-squamous, pem/cis (or carbo)+PDR001+canakinumab
Drug: Gemcitabine — Intravenous infusion
  Arms: Group A: squamous, gem/cis+PDR001
Drug: Pemetrexed — Intravenous infusion
  Arms: Group B: non-squamous, pem/cis+PDR001; Group E: non-squamous, pem/cis (or carbo)+PDR001+canakinumab
Drug: Carboplatin — Intravenous infusion
  Arms: Group C: paclitaxel/carbo+PDR001; Group E: non-squamous, pem/cis (or carbo)+PDR001+canakinumab
Drug: Paclitaxel — Intravenous infusion
  Arms: Group C: paclitaxel/carbo+PDR001
Drug: Canakinumab — Subcutaneous injection
  Arms: Group E: non-squamous, pem/cis (or carbo)+PDR001+canakinumab

SUMMARY:
The primary purpose of this study is to establish the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) of PDR001 when administered in combination with platinum-doublet chemotherapy and other immunooncology agent(s) in treatment naive patients with PD-L1 unselected, advanced NSCLC, and to estimate the preliminary anti-tumor activity in this patient population.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patient has stage IIIB (and is not a candidate for definitive multimodality therapy) or has stage IV NSCLC or relapsed locally advanced or metastatic NSCLC as follows:

   1. Group A, group B and group C only: Patients not previously treated with any systemic anti-cancer therapy (e.g. cytotoxic drugs, targeted therapy, monoclonal antibody therapy including immunotherapy (e.g. PD-1/PD-L1 inhibitors) or targeted therapies, either experimental or not), with exception of neo-adjuvant or adjuvant therapy as depicted in inclusion criterion 4.
   2. Group D only: Patients who have received only one prior systemic therapy treatment consisting of a PD-1 and/or PD-L1 inhibitor with or without a CTLA4 inhibitor for NSCLC, with exception of neo-adjuvant or adjuvant therapy as depicted in inclusion criterion 4. The last dose of prior immunotherapy must have been administered at least 6 weeks prior to the start of study treatment (cycle 1 day 1).
2. Histologically or cytologically confirmed diagnosis of NSCLC that is EGFR Wild-type, ALK-negative rearrangement and ROS1-negative rearrangement
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
4. Patients with at least 1 measurable tumor lesion as assessed by Computed Tomography (CT) Scan or Magnetic Resonance Imaging (MRI) according to RECIST 1.1.

Main Exclusion Criteria:

1. Patient with a history of severe hypersensitivity reaction to the planned study treatment including gemcitabine, paclitaxel, cisplatin, carboplatin, pemetrexed or any known excipients of these drugs
2. History of severe hypersensitivity reactions to other monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction.
3. Patient has history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic intervention).
4. History of leptomeningeal metastases
5. Active, known or suspected autoimmune disease or a documented history of autoimmune disease, including ulcerative colitis and Crohn's disease (Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll).
6. Use of any live vaccines against infectious diseases within 4 weeks of initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) during the first 6 weeks of therapy | 42 days
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 42 days
Overall response rate (ORR) per local investigator assessment for groups A, B and C | From baseline up to approximately 28 months
  ORR is defined as the proportion of patients with best overall response (BOR) of complete response (CR) or partial response (PR), as per RECIST 1.1 and local investigator assessment for groups A, B and C

SECONDARY OUTCOMES:
Overall Response Rate (ORR) per local investigator assessment for group E | Up to approximately 28 months
  ORR is defined as the proportion of patients with BOR of CR or PR, as per RECIST 1.1 and local investigator assessment for group E
Progression Free Survival (PFS) per Investigator | From start of treatment to the date of the first documented progression or death due to any cause, whichever comes first, assessed up to approximately 28 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause, as per RECIST 1.1 and local investigator assessment
Disease Control Rate (DCR) per Investigator | Up to approximately 28 months
  DCR is the proportion of patients with a BOR of CR or PR or stable disease (SD), as per RECIST 1.1 and local investigator assessment.
Duration of Response (DOR) per Investigator | From date of first documented response to the first documented progression or death due to any cause, whichever comes first, assessed up to approximately 28 months
  DOR is defined by responders as the time between the date of first documented response (CR or PR) and the date of first documented progression (RECIST 1.1 and local investigator assessment) or death due any cause
Time to Response (TTR) per Investigator | From start of treatment to the date of the first documented reponse (CR or PR), assessed up to approximately 28 months
  TTR is defined as the time from the date of start of treatment to the first documented response of either CR or PR as per RECIST 1.1 and local investigator assessment
Overall survival (OS) | from date of start of treatment to date of death due to any cause (assessed up to approximately 3.5 years)
  OS is defined as the time from date of start of treatment to date of death due to any cause.
Trough plasma Concentration (Ctrough) of PDR001 | Pre-infusion on Day 1 of Cycle 1 to 4 of induction phase; pre-infusion on Day 1 of Cycle 1 to 4, 6, 8 and every 6 cycle afterwards of maintenance phase; Cycle = 21 Days
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
Trough plasma Concentration (Ctrough) of chemotherapy | Pre-infusion on Day 1 of Cycle 1, 3 and 4 of induction phase; Cycle = 21 Days
  Blood samples will be collected at indicated time points for pharmacokinetic analysis. Ctrough will be assessed for all chemotherapy agents: cysplatin, pemetrexed, carboplatin and gemcitabine
Trough plasma Concentration (Ctrough) of canakinumab | Pre-infusion on Day 1 of Cycle 1, 3 and 4 of induction phase; Cycle = 21 Days
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
PDR001 Antidrug antibodies (ADA) prevalence at baseline | Baseline
  Blood samples will be collected at indicated time points for immunogenicity analysis.
Canakinumab ADA prevalence at baseline | Baseline
  Blood samples will be collected at indicated time points for immunogenicity analysis.
PDR001 ADA incidence during treatment | Pre-infusion on Day 1 of Cycle 1 to 4 of induction phase, pre-infusion on Day 1 of Cycle 1, 2, 3, 4, 6, 8 and every 6 cycle afterwards of maintenance phase, end of treatment and 30 and 150-day post-treatment
  Blood samples will be collected at indicated time points for immunogenicity analysis.
Canakinumab ADA incidence during treatment | Pre-infusion on Day 1 of Cycle 1 and 4 of induction phase, pre-infusion on Day 1 of Cycle 6, 14 and 20 of maintenance phase, end of treatment and 30 and 150-day post-treatment
  Blood samples will be collected at indicated time points for immunogenicity analysis.
Incidence of Adverse Events (AEs) | through study completion, up to approximately 3.5 years
  Incidence of AEs (CTCAE v4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (5):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - UCLA Santa Monica Hematology / Oncology SC-2, Santa Monica, California
  - Stanford Cancer Center SC, Stanford, California
  - Henry Ford Health System SC, Detroit, Michigan
  - Washington University School of Medicine SC, St Louis, Missouri
- Belgium (2):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Roeselare
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Prague, Czechia
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
- Germany (2):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Göttingen
- Novartis Investigative Site, Pokfulam, Hong Kong, Hong Kong
- Italy (3):
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Aviano, PN
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santoro A, Pilar G, Tan DSW, Zugazagoitia J, Shepherd FA, Bearz A, Barlesi F, Kim TM, Overbeck TR, Felip E, Cai C, Eddy S, McCulloch T, Schaefer ES. Spartalizumab in combination with platinum-doublet chemotherapy with or without canakinumab in patients with PD-L1-unselected, metastatic NSCLC. BMC Cancer. 2024 Oct 24;24(1):1307. doi: 10.1186/s12885-024-12841-2. PMID 39448966
- See also: Results for CPDR001C2101 from the Novartis Clinical Trial Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17963
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1108